CLINICAL TRIAL: NCT02402842
Title: Assessment of the Clinical Value of a Docetaxel, Cisplatin and 5-fluorouracil (DCF) Strategy Adapted to Patients for the Management of Metastatic or Locally Advanced Anal Resistant Radiochemotherapy Squamous Cell Anal Carcinoma.
Brief Title: Clinical and Biological Interest of Taxanes in Advanced Squamous Cell Anal Carcinoma
Acronym: Epitopes-HPV02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Epitopes-HPV02; 2014-001789-81 (EudraCT Number)
Record Dates: First submitted 2014-11-27; First posted 2015-03-30 (Estimated); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Anal Canal Carcinoma
Keywords: gastrointestinal oncology; immunology; taxane
MeSH Terms: conditions — Anal Canal Carcinoma | interventions — Docetaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DCF regimen (Experimental): docetaxel 75 mg/m2 day, Cisplatin75 mg/m2 and 5Fluorouracil at 750 mg/m2/day for 5 days
  Interventions: Drug: Docetaxel, Cisplatin and 5-Fluorouracil

INTERVENTIONS:
Drug: Docetaxel, Cisplatin and 5-Fluorouracil — Patients will receive 6 cycles of DCF regimen (docetaxel 75 mg/m2 day, cisplatin 75 mg/m2 and 5 Fluorouracil at 750 mg/m2/day for 5 days) every 3 weeks or 8 cycles of modified-DCF regimen (docetaxel 40 mg/m2 day, cisplatin 40 mg/m2 day and 5-Fluorouracil at 1200 mg/m2/day for 2 days) every 2 weeks, according to their clinical status.

SUMMARY:
Squamous cell carcinoma of the anal canal (SCCA) is a rare disease and mostly diagnosed at an early stage. After standard concurrent chemoradiation (CRT) with mitomycin (MMC) and 5-fluorouracil (5FU), the disease will recur in 20% of patients. After treatment failure (including salvage surgery), cisplatin-5FU combination is the standard option but complete response is a rare event and the prognosis remains poor with most patients' death occurring in the first 12 months. Decision making for physicians in this setting is only based on retrospective studies or small phase II clinical trials including less than 20 patients. Hence, no efficient standard of care is currently available for relapsing SCCA patients who are currently treated with a palliative intent.

Between 2007 and 2013, 8 consecutive patients with advanced recurrent SCCA after CRT were treated with DCF regimen (docetaxel, cisplatin and 5-fluorouracil) in the Regional Cancer Institute of Franche Comté. After a median follow-up of 41 months, 4 patients (50%) achieved a complete response. Three patients underwent surgery of all involved metastatic sites. A pathological complete response was observed for all of them including in metastases occurring in irradiated fields, suggesting that taxane-based chemotherapy might be an effective strategy to circumvent resistance to radiotherapy (a preliminary cohort of 8 patients was published (Kim S et al Annals of oncology 2013). Furthermore, all complete responders were HPV 16, and high levels of specific T cell responses against Human Papillomavirus (HPV) HPV16-derived E6/E7 and telomerase were detected in 50% of complete responders suggesting the potential restoration of cancer immunosurveillance by this regimen.

Then, the Epitopes-HPV02 multicenter phase II study will aim to confirm the new role of taxane-based chemotherapy in SCCA patients.

DETAILED DESCRIPTION:
Epitopes-HPV02 study is a national multicenter open label phase II trial including 66 patients.

Patients will receive 6 cycles of DCF regimen (docetaxel 75 mg/m2 day, CDDP 75 mg/m2 and 5FU at 750 mg/m2/day for 5 days) every 3 weeks or 8 cycles of modified-DCF regimen (docetaxel 40 mg/m2 day, CDDP 40 mg/m2 day and 5-FU at 1200 mg/m2/day for 2 days) every 2 weeks, according to their clinical status.

CT scan will be planned at baseline, after 3 and after 6 cycles of DCF regimen (or after 4 and 8 cycles of modified-DCF regimen) and then every three months until disease progression or death. A Pet-scan will be performed before and after 6 cycles of DCF. Tumor assessment will be carried out according to RECIST V1.1 criteria.

This study is carried out by the University Hospital of Besançon and were approved by the independent Est-II French Committee for Protection of Persons (CPP) and by the French Health Products Safety Agency (ANSM). This study will be conducted in 17 clinical centers in France.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Performance status ECOG-WHO ≤ 1
* histologically proved and unresectable locally advanced or metastatic squamous cell anal carcinoma
* patient eligible to DCF regimen
* signed written informed consent

Exclusion Criteria:

* known hypersensitivity or contraindication to any of the study drugs (docetaxel, cisplatin, 5-fluorouracil).
* previous chemotherapy for metastatic disease
* previous chemotherapy by paclitaxel, docetaxel or navelbine
* previous chemotherapy by cisplatin, except of concomitant radiotherapy
* SIDA
* clinically significant cardiac disease
* other malignancy within the last 3 years, except for adequately treated carcinoma in situ of the cervix or squamous carcinoma of the skin, or adequately controlled limited basal cell skin cancer.
* simultaneous participation in another clinical study
* pregnancy, breast-feeding or absence of adequate contraception for fertile patients
* patient with any medical or psychiatric condition or disease which would make the patient inappropriate for entry into this study.
* patient under guardianship, curator or under the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-09; Primary Completion 2018-06 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate | 12 months after initiation of chemotherapy DCF.
  Progression-free survival observed = the number of patients alive without progression at 12 months.

SECONDARY OUTCOMES:
Overall survival | date of death from any cause (within 3 years after the initiation of the treatment)
  time between the date of initiation of treatment and the date of death from any cause.
Progression free survival | date of first progression of the disease (within 3 years after the initiation of the treatment)
  time interval between the date of initiation of treatment and the date of first progression (local, remote [extent of the disease by RECIST v1.1] second cancer) or death from any cause.
response rate | 4 weeks after the end of DCF regimen
  response rate will be evaluated using Response Evaluation Criteria in Solid Tumor (RECIST) v1.1 by CT-scan
Tolerance of the DCF regimen ( Common Terminology Criteria for Adverse Events version 4.03) | from the initiation of DCF regimen to 4 weeks after the end of DCF regimen
  description of toxicities and adverse events according to Common Terminology Criteria for Adverse Events version 4.03
quality of life related to health | from the inclusion to patient death or for maximum 3 years after end of treatment
  EORTC-QLQ-C30 & time to QoL score deterioration
HPV-specific T cell responses measured by ELISPOT assay before and after DCF treatment | at baseline (inclusion) and 4 weeks after the end of DCF regimen
  HPV-specific T cell responses measured by ELISPOT assay

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - University hospital of Besançon, Besançon
  - FNLCC center Georges François Leclerc, Dijon
  - Oscar Lambret center, Lille
  - Jean Mermoz Private Hospital, Lyon
  - Hospital of Belfort-Montbeliard, Montbéliard
  - Regional Institute of Cancer, Montpellier
  - Institute of Cancerology of Lorraine, Nancy
  - Antoine Lacassagne Center, Nice
  - Paris Saint-Joseph Hospital Group, Paris
  - Curie Institute, Paris
  - Pitié Salpétrière Hospital, Paris
  - Mutualist Montsouris Institute, Paris
  - European Georges Pompidou Hospital, Paris
  - Saint-Antoine Hospital, Paris
  - University Robert Debré Hospital, Reims
  - Paul Strauss Center, Strasbourg

REFERENCES:
- [Background] Kim S, Jary M, Mansi L, Benzidane B, Cazorla A, Demarchi M, Nguyen T, Kaliski A, Delabrousse E, Bonnetain F, Letondal P, Bosset JF, Valmary-Degano S, Borg C. DCF (docetaxel, cisplatin and 5-fluorouracil) chemotherapy is a promising treatment for recurrent advanced squamous cell anal carcinoma. Ann Oncol. 2013 Dec;24(12):3045-50. doi: 10.1093/annonc/mdt396. Epub 2013 Oct 10. PMID 24114858
- [Background] Kim S, Meurisse A, Spehner L, Stouvenot M, Francois E, Buecher B, Andre T, Samalin E, Jary M, Nguyen T, El Hajbi F, Baba-Hamed N, Pernot S, Kaminsky MC, Bouche O, Desrame J, Zoubir M, Ghiringhelli F, Parzy A, de la Fouchardiere C, Boulbair F, Lakkis Z, Klajer E, Jacquin M, Taieb J, Vendrely V, Vernerey D, Borg C. Pooled analysis of 115 patients from updated data of Epitopes-HPV01 and Epitopes-HPV02 studies in first-line advanced anal squamous cell carcinoma. Ther Adv Med Oncol. 2020 Dec 4;12:1758835920975356. doi: 10.1177/1758835920975356. eCollection 2020. PMID 33329760
- [Background] Spehner L, Kim S, Vienot A, Francois E, Buecher B, Adotevi O, Vernerey D, Abdeljaoued S, Meurisse A, Borg C. Anti-Telomerase CD4+ Th1 Immunity and Monocytic-Myeloid-Derived-Suppressor Cells Are Associated with Long-Term Efficacy Achieved by Docetaxel, Cisplatin, and 5-Fluorouracil (DCF) in Advanced Anal Squamous Cell Carcinoma: Translational Study of Epitopes-HPV01 and 02 Trials. Int J Mol Sci. 2020 Sep 17;21(18):6838. doi: 10.3390/ijms21186838. PMID 32957741
- [Background] Stouvenot M, Meurisse A, Saint A, Buecher B, Andre T, Samalin E, Jary M, El Hajbi F, Baba-Hamed N, Pernot S, Kaminsky MC, Bouche O, Desrame J, Zoubir M, Smith D, Ghiringhelli F, Parzy A, de la Fouchardiere C, Almotlak H, Vienot A, Jacquin M, Taieb J, Nguyen T, Vernerey D, Borg C, Kim S. Second-line treatment after docetaxel, cisplatin and 5-fluorouracil in metastatic squamous cell carcinomas of the anus. Pooled analysis of prospective Epitopes-HPV01 and Epitopes-HPV02 studies. Eur J Cancer. 2022 Feb;162:138-147. doi: 10.1016/j.ejca.2021.11.019. Epub 2022 Jan 4. PMID 34995900
- [Result] Kim S, Francois E, Andre T, Samalin E, Jary M, El Hajbi F, Baba-Hamed N, Pernot S, Kaminsky MC, Bouche O, Desrame J, Zoubir M, Ghiringhelli F, Parzy A, De La Fouchardiere C, Smith D, Deberne M, Spehner L, Badet N, Adotevi O, Anota A, Meurisse A, Vernerey D, Taieb J, Vendrely V, Buecher B, Borg C. Docetaxel, cisplatin, and fluorouracil chemotherapy for metastatic or unresectable locally recurrent anal squamous cell carcinoma (Epitopes-HPV02): a multicentre, single-arm, phase 2 study. Lancet Oncol. 2018 Aug;19(8):1094-1106. doi: 10.1016/S1470-2045(18)30321-8. Epub 2018 Jul 2. PMID 30042063
- [Derived] Kim S, Jary M, Andre T, Vendrely V, Buecher B, Francois E, Bidard FC, Dumont S, Samalin E, Peiffert D, Pernot S, Baba-Hamed N, El Hajbi F, Bouche O, Desrame J, Parzy A, Zoubir M, Louvet C, Bachet JB, Nguyen T, Abdelghani MB, Smith D, De La Fouchardiere C, Aparicio T, Bennouna J, Gornet JM, Jacquin M, Bonnetain F, Borg C. Docetaxel, Cisplatin, and 5-fluorouracil (DCF) chemotherapy in the treatment of metastatic or unresectable locally recurrent anal squamous cell carcinoma: a phase II study of French interdisciplinary GERCOR and FFCD groups (Epitopes-HPV02 study). BMC Cancer. 2017 Aug 25;17(1):574. doi: 10.1186/s12885-017-3566-0. PMID 28841909